CLINICAL TRIAL: NCT05223075
Title: Articaine Versus Lidocaine in Only Buccal Infiltration Anesthesia for the Extraction of Mandibular Anterior Teeth.Asplit Mouth Clinical Trail
Brief Title: Articaine Versus Lidocaine Buccal Infiltration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofaciall surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 256-06/2018
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pain
Keywords: buccal infiltration; lidocaine; articaine
MeSH Terms: conditions — Pain | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- articaine group (Experimental)
  Interventions: Drug: articaine local anethesia with vasoconstrictor
- lidocaine group (Experimental)
  Interventions: Drug: lidocaine local anethesia with vasoconstrictor

INTERVENTIONS:
Drug: articaine local anethesia with vasoconstrictor — buccal infiltration only of articaine local anethesia during extraction of lower anterior teeth
  Arms: articaine group
Drug: lidocaine local anethesia with vasoconstrictor — buccal infiltration only of lidocaine local anethesia during extraction of lower anterior teeth
  Arms: lidocaine group

SUMMARY:
assess the effect of articaine versus lidocaine in only buccal infiltration of local anethesia in lower anterior teeth

ELIGIBILITY:
Inclusion Criteria:

* medically stable
* 18years or older
* patient with bilateral lower anterior teeth requiring non surgical removal

Exclusion Criteria:

* grade 3 mobility
* neurological disease
* allergy to anethesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
pain during extraction | during extraction
  by (VAS) visual analouge scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

REFERENCES:
- [Derived] Al-Mahalawy H, El-Mahallawy Y, Abdelrahman HH, Refahee SM. Articaine versus Lidocaine in only buccal infiltration anesthesia for the extraction of mandibular anterior teeth. A prospective split-mouth randomized-controlled clinical study. BMC Oral Health. 2023 Aug 28;23(1):604. doi: 10.1186/s12903-023-03292-5. PMID 37641122